CLINICAL TRIAL: NCT07050160
Title: A Phase 1/2 Long-term Follow-up Study of the Safety and Efficacy of LX2020 Gene Therapy in Patients With Arrhythmogenic Cardiomyopathy Due to a Plakophilin-2 Pathogenic Variant
Brief Title: Long-term Follow-up Study of Gene Therapy for Arrhythmogenic Cardiomyopathy Due to a Plakophilin-2 Pathogenic Variant
Acronym: GRIT-PKP2
Status: Enrolling by invitation | Type: Observational
Sponsor: Lexeo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: LX2020-02
Record Dates: First submitted 2025-06-11; First posted 2025-07-03 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Arrhythmogenic Cardiomyopathy; PKP2-ACM; PKP2-ARVC
Keywords: Arrhythmogenic Cardiomyopathy; ACM; Cardiomyopathy; ARVC; Arrhythmogenic Right Ventricular; Arrhythmogenic Right Ventricular Dysplasia; Genetic cardiomyopathy; Gene Therapy; PKP2 Gene; Plakophilin-2; LX2020; GRIT-PKP2; Ventricular Arrhythmia; PVCs; Sudden Cardiac Death; Cardiac Arrest
MeSH Terms: conditions — Cardiomyopathies; Arrhythmogenic Right Ventricular Dysplasia; Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LX2020 treated participants: Participants who received LX2020 in Study LX2020-01

SUMMARY:
The primary objective of this Phase 1/2 long-term follow-up (LTFU) study is to assess the long-term safety and tolerability of LX2020 for the treatment of arrhythmogenic cardiomyopathy (ACM) due to a plakophilin-2 gene (PKP2) pathogenic variant (PKP2-ACM).

DETAILED DESCRIPTION:
GRIT-PKP2 is a Phase 1/2 long-term follow-up (LTFU) study designed to evaluate the long-term safety and tolerability of LX2020 gene therapy for participants with PKP2-ACM who have previously received LX2020 in the parent study, LX2020-01. After completion of Study LX2020-01, participants will roll over into this study LX2020-02 for an additional 4-year long-term observation. No gene therapy will be administered in Study LX2020-02. Efficacy will be assessed as an exploratory objective.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received LX2020 in study LX2020-01

Exclusion Criteria:

* Concurrent enrollment in any other clinical investigation involving use of an investigational agent.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received LX2020 in Study LX2020-01 will roll over into this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who experienced at least 1 treatment emergent adverse event (TEAE) and/or 1 treatment emergent serious adverse event (TESAE). | 4 years
  Evaluation of Safety and Tolerability of LX2020

OTHER OUTCOMES:
Selected Exploratory | 4 years
  Change in the frequency of ventricular arrhythmias from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lexeo Clinical Trials, Study Director — Lexeo Therapeutics
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States